CLINICAL TRIAL: NCT05859659
Title: Clinical, patHOlogical and Imaging Project of nEuro-oncology (HOPE)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yaou Liu, Professor, Beijing Tiantan Hospital
Other Study IDs: KY2022-078-04
Record Dates: First submitted 2023-05-05; First posted 2023-05-16 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Molecular pathology of glioma positive
  Interventions: Diagnostic Test: This study does not intervene in this process.
- Molecular pathology of glioma negative
  Interventions: Diagnostic Test: This study does not intervene in this process.

INTERVENTIONS:
Diagnostic Test: This study does not intervene in this process. — This study does not intervene in this process.

SUMMARY:
Glioma disease is the most common primary malignant tumor of the central nervous system, with an annual incidence of about 3-8 people per 100,000 population, of which glioblastoma with the highest degree of malignancy and the worst prognosis accounts for 70-75%. The construction goal of this project is to construct a multivariate retrospective glioma database (3000 cases) integrating clinical information, magnetic resonance imaging examination and molecular pathological results, and a prospective glioma database (500 cases) integrating advanced magnetic resonance sequences. It aims to form a standardized database integrating clinical-prognostic information, magnetic resonance imaging and pathological results. Based on the construction of the above standardized database, the specifications for the acquisition of cranial magnetic resonance images, the image segmentation and labeling process, and the expert consensus on database construction and use management of glioma diseases were established. Form a multimodal, large-capacity, high-quality, and rich medical imaging database that conforms to the characteristics of Chinese groups and clinical diagnosis and treatment norms; On this basis, the data are dynamically updated, in-depth mining, and the classification and grading standards of glioma diseases, prognosis judgment criteria and treatment efficacy evaluation system are formulated.

DETAILED DESCRIPTION:
Glioma disease is the most common primary malignant tumor of the central nervous system, with an annual incidence of about 3-8 people per 100,000 population, of which glioblastoma with the highest degree of malignancy and the worst prognosis accounts for 70-75%. The construction goal of this project is to construct a multivariate retrospective glioma database (3000 cases) integrating clinical information, magnetic resonance imaging examination and molecular pathological results, and a prospective glioma database (500 cases) integrating advanced magnetic resonance sequences. It aims to form a standardized database integrating clinical-prognostic information, magnetic resonance imaging and pathological results. Based on the construction of the above standardized database, the specifications for the acquisition of cranial magnetic resonance images, the image segmentation and labeling process, and the expert consensus on database construction and use management of glioma diseases were established. Form a multimodal, large-capacity, high-quality, and rich medical imaging database that conforms to the characteristics of Chinese groups and clinical diagnosis and treatment norms; On this basis, the data are dynamically updated, in-depth mining, and the classification and grading standards of glioma diseases, prognosis judgment criteria and treatment efficacy evaluation system are formulated.

ELIGIBILITY:
Inclusion Criteria:

* (1) a clear diagnosis of glioma based on pathological results;
* (2) The MRI sequence is complete and there are no obvious artifacts in the image;
* (3) The patient signs an informed consent form

Exclusion Criteria:

* (1) Suffering from other neurological diseases;
* (2) Prior to enrollment, surgery or biopsy, or a history of radiation therapy or chemotherapy;
* (3) Unable to complete clinical scoring and related laboratory tests, unable to complete follow-up;
* (4) Unable to tolerate MRI examination; Poor image quality, such as motion artifacts.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: To reflect the daily practices, this study includes all patients with diffuse glioma at the beginning of the study.
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Establish standardized clinical-MRI -molecular markers database for glioma | 2022.01-2024.12
  1) Collect clinical, MRI and molecular markers data of glioma patients; 2) Establish a standardized tumor labeling database; 3) Establish an automatic segmentation and recognition model of glioma
Establish an accurate MRI-based deep-learning model for the prediction of glioma | 2022.01-2024.12
  1) Build an accurate MRI-based deep-learning model with retrospective data. 2) The multicenter data was used to verify the repeatability and widespread use of the model again

CONTACTS AND LOCATIONS:
Overall Officials: Yaou Liu, Doctor, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Clinical and MR data can be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 3 years after the end of the trial.
Access Criteria: Neurosurgeon and radiologist who submitting an application to Prof. Liu.